CLINICAL TRIAL: NCT03129048
Title: Mediterranean Diet, Weight Loss, and Cognition in Obese Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dr. Fitzgibbon, Professor Department of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-0258
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cognition; Obese Older Adults; Mediterranean Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MedDiet-WL (Experimental): MedDiet-WL group, advice and exchange lists will be designed to promote a 1-2 lb. per week weight loss (approximately 30% caloric restriction or a reduction of about 600 calories per day) for an end goal of a 7% weight loss from baseline.
  Interventions: Behavioral: MedDiet
- MedDiet-A (Experimental): For the MedDiet-A group, dietary advice and corresponding exchange lists will be given within the context of promoting weight stability.
  Interventions: Behavioral: MedDiet
- Typical Diet Control (TDC) (Other): Typical Diet Control (TDC) will maintain current eating and activity patterns and weight over 14 months.
  Interventions: Behavioral: MedDiet

INTERVENTIONS:
Behavioral: MedDiet — Research subjects will be randomly assigned to one of three intervention groups.
  The MedDiet-A group will learn about and how to adhere to the Mediterranean Diet. Over the course of 8 months, they will receive twenty-two classes 60-minute in length.
  The MedDiet-WL group will learn about the Mediterranean Diet, how to adhere to is and engage in lifestyle choices like exercising and eating fewer calories so that they will loose weight. Over the course of 8 months they will receive 22 classes, each 90 minutes in length.
  The Typical Diet Control group will be asked to maintain current eating and activity patterns over the course of the 14 month study.

SUMMARY:
The deleterious effects of obesity on cardiovascular disease (CVD) and metabolic risk factors (dyslipidemia, hypertension, and insulin resistance) are well-documented. Recent evidence also links obesity to cognitive decline and dementia. Dietary patterns are central to the development and maintenance of obesity and certain dietary patterns may contribute to the onset and progression of cognitive decline. With the rapid aging of the US population and the high prevalence of obesity among older adults, innovative lifestyle strategies to prevent cognitive decline among ethnically diverse obese older adults are critically needed.

DETAILED DESCRIPTION:
Obesity is a leading cause of death and disability in the United States, affecting as many as 80 million Americans. It is well-established that obesity contributes to a number of risk factors for metabolic abnormalities and cardiovascular diseases (CVD), including hypertension, diabetes, and hyperlipidemia. In addition, there is growing evidence that obesity is associated with cognitive deficits in multiple domains, even in otherwise healthy older adults. With the rapidly aging US population and the high prevalence of obesity among older adults, innovative strategies to prevent cognitive decline in this population are needed. Dietary patterns are central to the development and maintenance of obesity and evidence suggests that dietary factors also may affect cognition. Studies have shown that adherence to a Mediterranean Diet (MedDiet) is associated with less cognitive decline and reduced risk for dementia in older adults. Weight loss through caloric restriction also has been shown to improve cognitive function in obese adults. Both the MedDiet and weight loss are thought to improve cognition in obese individuals and reduce CVD/metabolic risk through beneficial changes in systemic inflammation and oxidative stress. The identification of effective lifestyle interventions for diet/weight management to improve cognition among obese older adults is a public health priority. However, no randomized controlled trials (RCTs) have examined the effect of the MedDiet with and without caloric restriction, to promote weight loss on cognitive functioning in obese older adults. The investigators propose a three-arm RCT in which 180 obese (body mass index [BMI] ≥ 30 and < 50 kg/m²) older adults (55-80 years) will be randomized to: 1) an 8-month MedDiet Alone, without caloric restriction/weight loss (MedDiet-A); 2) an 8-month MedDiet lifestyle intervention with caloric restriction/weight loss (MedDiet-WL); or 3) an 8-month typical diet control (TDC) without caloric restriction/weight loss. The investigators will test the following hypotheses: 1) participants randomized to MedDiet-A and MedDiet-WL will achieve greater improvements in cognition compared to participants randomized to TDC; 2) participants randomized to MedDiet-WL will exhibit greater improvements in cognition compared to participants randomized to MedDiet-A; 3) participants randomized to MedDiet-A and MedDiet-WL will show greater improvements in CVD/metabolic risk factors, systemic inflammation, OxStress, and body weight/composition compared to participants in TDC; 4) participants randomized to MedDiet-WL will exhibit greater improvements in CVD/metabolic risk factors, systemic inflammation, OxStress, and body weight/composition compared to MedDiet-A; 5) improvements in CVD/metabolic risk factors, body composition, systemic inflammation, and OxStress will mediate the relationship between MedDiet and improved cognition. The investigators also will determine the extent to which changes in dietary habits, weight and cognitive functioning are maintained over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 55 years of age],
* BMI 30.0-50.0 kg/m2,
* English speaking
* Have access to a phone
* Plan to reside in the Chicago area for the following 14 months
* Minimal levels of cognitive impairment as determined by the Montreal Cognitive Assessment (MoCA) < 19.

Exclusion Criteria:

* The exclusion criteria ensure that participants can safely participate in the trial.
* renal disease
* autoimmune disorder
* immunodeficiency
* malabsorptive disorder
* gastrointestinal and hepatic diseases
* severe ischemic heart disease
* severe pulmonary disease
* bariatric surgery
* alcohol abuse (> 50 grams/day) or illicit drug abuse
* uncontrolled diabetes based on capillary hemoglobin A1c (HbA1c) > 9.0%
* schizophrenia or bipolar disorder
* cancer treatment within the past 12 months
* weight > 450 lbs. (due to the weight limitation of the DXA scanner)
* diagnosed sleep apnea and regularly using a cpap machine
* currently adhering to a MedDiet, Montreal Cognitive Assessment (MoCA) < 19,(161) -
* currently on a weight-loss diet or actively involved in a formal weight loss program (e.g., Weight Watchers.)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Assessing change in Attention between time periods | 14 months
  Baseline, 8-month (first intervention), and 14-month assessments will include Digit Symbol test.
Assessing change in Executive Function between time periods | 14 months
  Baseline, 8-month (first intervention), and 14-month assessments will include the Trail Making Test Part B.
Assessing change in Memory between time periods | 14 months
  Baseline, 8-month (first intervention), and 14-month assessments will include tests of memory including the delayed free recall from the Hopkins Verbal Learning Test.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Fitzgibbon, PhD, Principal Investigator — UIC
Locations (1):
- University Of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fitzgibbon M, Blumstein L, Schiffer L, Antonic MA, McLeod A, Dakers R, Restrepo L, Boots EA, Sanchez-Flack JC, Tussing-Humphreys L, Lamar M. Adapting to the COVID-19 pandemic on Building Research in Diet and Cognition (BRIDGE) trial. Trials. 2021 Jul 16;22(1):459. doi: 10.1186/s13063-021-05383-6. PMID 34271944
- [Derived] Fitzgibbon M, Blumstein L, Schiffer L, Antonic MA, McLeod A, Dakers R, Restrepo L, Boots EA, Sanchez-Flack JC, Tussing-Humphreys L, Lamar M. Adapting to the impact of the COVID-19 pandemic on a randomized controlled trial examining lifestyle behaviors on cognitive functioning in obese African American adults: Building Research in Diet and Cognition (BRIDGE). Res Sq [Preprint]. 2021 Apr 26:rs.3.rs-290482. doi: 10.21203/rs.3.rs-290482/v1. PMID 34013252